CLINICAL TRIAL: NCT03840850
Title: Type 2 Diabetes: Risk Perceptions and Self-management Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: NIHR Collaboration for Leadership in Applied Health Research and Care (Oxford) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17/NW/0267
Record Dates: First submitted 2019-01-18; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention and usual care (Experimental): Risk communication intervention and usual care including personalized lifestyle advice
  Interventions: Other: Personalized Risk Communication for People with Type 2 Diabetes
- Usual care only (No Intervention): Usual care including personalized lifestyle advice

INTERVENTIONS:
Other: Personalized Risk Communication for People with Type 2 Diabetes — The risk communication intervention consists of communicating the impact of being poorly controlled on two types of outcome: (1) absolute 10-year risk of experiencing a cardiovascular event, i.e. heart attack or stroke (10-year CV risk); (2) life expectancy. These personalized risk estimates are calculated based on the UKPDS outcomes model (version 2), which is a prognostic model of reference in the area of Type 2 diabetes.
  Arms: Intervention and usual care

SUMMARY:
This pilot randomised controlled trial (RCT) aims to assess the feasibility of using a new type of risk communication intervention for people with Type 2 diabetes mellitus (T2DM) in primary care and to evaluate its potential impact on risk perceptions and self-management behaviour.

The study comprises 40 participants with T2DM randomly allocated to usual care supported by the risk communication intervention or usual care only.

DETAILED DESCRIPTION:
Diabetes self-management, which includes self-care behaviours such as healthy eating and physical exercise, has become the cornerstone for treating type-2 diabetes mellitus (T2DM). However, although self-management education (SME) is necessary to equip patients with the knowledge, skills and attitudes required to manage their diabetes care, the most effective method to do so is still unclear.

Recent studies have shown that people with T2DM underestimated their risks of developing complications. Although behavioural processes are complex, wrong risk perceptions are a major impediment to the adoption of self-care behaviours and, as a result, an additional risk for the occurrence of adverse outcomes.

Existing risk communication interventions have shown mixed results, with many participants barely understanding the explanations of health professionals about risks and having poor recall of risk information. In this context, there is a need for better risk communication interventions.

Based on the results of recent studies investigating the risk perceptions and risk attitudes of people with T2DM, we have developed a new, tailored risk communication intervention. The objectives of this intervention are:

* To increase the awareness of risks for complications associated with type 2 diabetes.
* To encourage the adoption of recommended self-care behaviours.

The intervention has been developed in collaboration with both health professionals and patients. We have designed a pilot study to assess the feasibility of using the intervention in primary care and to evaluate its potential impact on patients' risk perceptions and self-management behaviour, in order to inform the design of a largest study (RCT to be conducted in the future)

The intervention lasts 5 minutes on average, conducted by the general practitioner (GP) during patients' routine primary care consultation. The study involves 40 participants with T2DM randomly allocated to usual care supported by the risk communication intervention or usual care only.

The research is supported by the National Institute for Health Research (NIHR) Collaboration for Leadership in Applied Health Research and Care Oxford at Oxford Health NHS Foundation Trust.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Diagnosed with type-2 diabetes.

Exclusion Criteria:

* Unable to provide informed consent.
* Non-English speaker.
* Not suitable for the study according to GP.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing the intervention in primary care: Binary outcome (feasible / not feasible), as judged by the investigators | 3 months
  Binary outcome (feasible / not feasible), as judged by the investigators following analysis of study pre-specified outcome measures.

SECONDARY OUTCOMES:
Recall of personalised risk information | 3 months
  Recall of personalised risk information is measured immediately and 3 months after the intervention.
  Type of question used: "The doctor has recently calculated your personalised risk information on his computer. Do you remember these numbers?
  Binary outcome: information recalled or information not recalled. Recall of information represents a better outcome. Rates of information recall (%) are compared between the two groups.
Intentions to make lifestyle changes | 3 months
  Intentions to make lifestyle changes are measured immediately before and after the intervention using the validated Determinants of Lifestyle Behaviour Questionnaire (DLBQ). The DLBQ consists of three parts: intentions to eat healthier, to increase physical activity, and to reduce smoking consumption. Intentions are assessed by a 5-point Likert scale ranging from 0 (strongly disagree) to 5 (strongly agree). Each dimension score is assessed individually. Higher scores represent a better outcome.
Change in self-management behaviour | 3 months
  Change in self-management behaviour from baseline to 3 months is measured using the validated Summary of Diabetes Self-Care Activities (SDSCA) questionnaire. This instrument explores six dimensions of self-management (healthy eating, physical activity, medication adherence, self-monitoring of blood glucose, foot checks and smoking behaviour), using the self-reported frequency of completing recommended activities during the past seven days as an outcome (SDSCA score ranging from 0 to 7 for each dimension). Each dimension score is assessed individually. Higher scores represent a better outcome.

OTHER OUTCOMES:
Consent rate | 3 months
  Rate of eligible subjects consenting to participate in the study (%)
Acceptability of the intervention | Immediately after the intervention
  Participants' acceptability of the intervention is measured using adapted questions from the COMRADE (Combined Outcome Measure for Risk communication And treatment Decision-making Effectiveness) scale, which was validated for use in the UK. This scale consists of 10 questions on a 5-point scale ranging from 0 (strongly disagree) to 5 (strongly agree) and is used immediately after the intervention. The scores of each question are combined to compute an average score. Higher average scores represent a better outcome.
Anxiety due to the intervention | Immediately after the inervention
  Following Welschen et al. (2012), a question adapted from Claassen et al. (2010) is used to assess how anxious participants are about their personalised risk information (7-point Likert scale ranging from 0 (not anxious at all) to 7 (very much anxious). Higher scores represent a worse outcome.
Worry due to the intervention | Immediately after the intervention
  Following Welschen et al. (2012), a question adapted from Claassen et al. (2010) is used to assess how worried participants are about their personalised risk information (7-point Likert scale ranging from 0 (not worried at all) to 7 (very much worried). Higher scores represent a worse outcome.
Retention rate | 3 months
  Rate of participants who stay enrolled in the study until it ends (%)
Rate of missing data | 3 months
  Rate of missing data in participants' self-reported questionnaires (%)

CONTACTS AND LOCATIONS:
Locations (1):
- 27 Beaumont Street Surgery Practice, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT03840850/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT03840850/ICF_001.pdf